CLINICAL TRIAL: NCT04616612
Title: Medication Adherence Given Individual SystemCHANGE(TM) in Advancing Nephropathy (MAGICIAN) Pilot Study
Acronym: MAGICIAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Rebecca Jane Ellis, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2001957718; R21NR019348-02 (NIH)
Record Dates: First submitted 2020-09-17; First posted 2020-11-05 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease(CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Two-group, randomized, controlled trial
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SystemCHANGE (TM) (Experimental): SystemCHANGE™ focuses on using patients' already established and reliable systems to support medication-taking, rather than focusing on personal effort and "remembering."When applied to medication adherence, the goal is to reduce medication-taking variability and move towards consistently taking medication with a 6-hour window of time (for daily medications like RAAS) and avoid missing medications. SystemCHANGE™ improvement cycles rely on efficient use of performance feedback in order to make decisions about whether system solutions work or if there is a need to select other solutions.
  Interventions: Behavioral: SystemCHANGE (TM)
- Attention Control (Active Comparator): Participants in the attention control will receive educational materials about chronic kidney disease (CKD). The content will be focused on diet, exercise, and living with CKD.
  Interventions: Other: Attention Control

INTERVENTIONS:
Behavioral: SystemCHANGE (TM) — Participants randomized to the refined SystemCHANGE™ intervention will receive 7 personalized sessions with a nurse-interventionist (session 1 virtual face-to-face, sessions 2-7 via phone) and weekly feedback MMS message reports delivered to mobile phones.
  Arms: SystemCHANGE (TM)
Other: Attention Control — Participants randomized to attention control will receive nurse-led kidney disease self-care education based on materials developed by The National Institute of Diabetes and Digestive and Kidney Diseases and The National Kidney Foundation. Similar to the intervention, participants will receive one virtual visit from the nurse-interventionist and 6 phone calls (weeks 2, 3, 4, 5, 6 and 7) and weekly educational MMS messages delivered by mobile phone.
  Arms: Attention Control

SUMMARY:
The purpose of this 2-group, randomized, controlled trial is to evaluate the refined SystemCHANGE™ against attention control patient education in CKD patients taking RAAS medications.

DETAILED DESCRIPTION:
In this study, the investigators will test a refined SystemCHANGE™ in patients taking RAAS inhibiting medications. Participants will be recruited from two sources: 1) the largest and most comprehensive health care system in the state and 2) one of the largest essential health care systems in the country. Data are collected at baseline, 8 weeks (immediately post-intervention), and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* prescribed at least 1 daily RAAS inhibiting medication
* CKD diagnosis estimated glomerular filtration rate (eGFR) category G1 to G4
* RAAS inhibiting medication adherence of <.85 documented during the screening phase
* proteinuria defined as a urine Protein-to-Creatinine ratio > 150 mg/g or urine Albumin-to-Creatinine ratio >30mg/g
* able to speak, hear, and understand English determined by the ability to participate and comprehend conversation about potential inclusion in the study
* self-reported ability to open a pill cap
* able to self-administer RAAS inhibiting medications
* willing to use a study phone
* has no cognitive impairment as determined by a score of 4 or greater on the 6-item Telephone Mental Status Screen Derived from the Mini-Mental Status Exam (cognitive screener)
* has no other diagnoses that may shorten life span, such as metastatic cancer
* is not currently hospitalized
* receives care through two approved health care systems

Exclusion Criteria:

* Participants with kidney failure defined by GFR <15 mL/min/1.73
* Participants will be excluded if they are receiving dialysis or have dialysis access placed (e.g. graft or arteriovenous fistula) in anticipation of starting dialysis.
* Kidney and kidney-pancreas transplant recipients will be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J. Ellis, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Nursing, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Tangkiatkumjai M, Walker DM, Praditpornsilpa K, Boardman H. Association between medication adherence and clinical outcomes in patients with chronic kidney disease: a prospective cohort study. Clin Exp Nephrol. 2017 Jun;21(3):504-512. doi: 10.1007/s10157-016-1312-6. Epub 2016 Jul 20. PMID 27438073
- [Background] Muntner P, Judd SE, Krousel-Wood M, McClellan WM, Safford MM. Low medication adherence and hypertension control among adults with CKD: data from the REGARDS (Reasons for Geographic and Racial Differences in Stroke) Study. Am J Kidney Dis. 2010 Sep;56(3):447-57. doi: 10.1053/j.ajkd.2010.02.348. Epub 2010 May 14. PMID 20471734
- [Background] Cedillo-Couvert EA, Ricardo AC, Chen J, Cohan J, Fischer MJ, Krousel-Wood M, Kusek JW, Lederer S, Lustigova E, Ojo A, Porter AC, Sharp LK, Sondheimer J, Diamantidis C, Wang X, Roy J, Lash JP; CRIC Study Investigators. Self-reported Medication Adherence and CKD Progression. Kidney Int Rep. 2018 Feb 2;3(3):645-651. doi: 10.1016/j.ekir.2018.01.007. eCollection 2018 May. PMID 29854972
- [Background] Williams A, Manias E, Walker R, Gorelik A. A multifactorial intervention to improve blood pressure control in co-existing diabetes and kidney disease: a feasibility randomized controlled trial. J Adv Nurs. 2012 Nov;68(11):2515-25. doi: 10.1111/j.1365-2648.2012.05950.x. Epub 2012 Feb 15. PMID 22335395
- [Background] Ong SW, Jassal SV, Miller JA, Porter EC, Cafazzo JA, Seto E, Thorpe KE, Logan AG. Integrating a Smartphone-Based Self-Management System into Usual Care of Advanced CKD. Clin J Am Soc Nephrol. 2016 Jun 6;11(6):1054-1062. doi: 10.2215/CJN.10681015. Epub 2016 May 12. PMID 27173169
- [Background] Conn VS, Ruppar TM, Enriquez M, Cooper P. Medication adherence interventions that target subjects with adherence problems: Systematic review and meta-analysis. Res Social Adm Pharm. 2016 Mar-Apr;12(2):218-46. doi: 10.1016/j.sapharm.2015.06.001. Epub 2015 Jun 15. PMID 26164400
- [Background] Easthall C, Song F, Bhattacharya D. A meta-analysis of cognitive-based behaviour change techniques as interventions to improve medication adherence. BMJ Open. 2013 Aug 9;3(8):e002749. doi: 10.1136/bmjopen-2013-002749. PMID 23935093
- [Background] Haynes RB, Ackloo E, Sahota N, McDonald HP, Yao X. Interventions for enhancing medication adherence. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD000011. doi: 10.1002/14651858.CD000011.pub3. PMID 18425859
- [Background] Ivers NM, Grimshaw JM, Jamtvedt G, Flottorp S, O'Brien MA, French SD, Young J, Odgaard-Jensen J. Growing literature, stagnant science? Systematic review, meta-regression and cumulative analysis of audit and feedback interventions in health care. J Gen Intern Med. 2014 Nov;29(11):1534-41. doi: 10.1007/s11606-014-2913-y. PMID 24965281
- [Background] Rambod M, Heine GH, Seiler S, Dominic EA, Rogacev KS, Dwivedi R, Ramezani A, Wing MR, Amdur RL, Fliser D, Raj DS. Association of vascular endothelial factors with cardiovascular outcome and mortality in chronic kidney disease patients: a 4-year cohort study. Atherosclerosis. 2014 Oct;236(2):360-5. doi: 10.1016/j.atherosclerosis.2014.07.026. Epub 2014 Aug 12. PMID 25128974
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Debella YT, Giduma HD, Light RP, Agarwal R. Chronic kidney disease as a coronary disease equivalent--a comparison with diabetes over a decade. Clin J Am Soc Nephrol. 2011 Jun;6(6):1385-92. doi: 10.2215/CJN.10271110. Epub 2011 Mar 10. PMID 21393492
- [Background] Jafar TH, Stark PC, Schmid CH, Landa M, Maschio G, de Jong PE, de Zeeuw D, Shahinfar S, Toto R, Levey AS; AIPRD Study Group. Progression of chronic kidney disease: the role of blood pressure control, proteinuria, and angiotensin-converting enzyme inhibition: a patient-level meta-analysis. Ann Intern Med. 2003 Aug 19;139(4):244-52. doi: 10.7326/0003-4819-139-4-200308190-00006. PMID 12965979
- [Background] Evans M, Bain SC, Hogan S, Bilous RW; Collaborative Study Group participants. Irbesartan delays progression of nephropathy as measured by estimated glomerular filtration rate: post hoc analysis of the Irbesartan Diabetic Nephropathy Trial. Nephrol Dial Transplant. 2012 Jun;27(6):2255-63. doi: 10.1093/ndt/gfr696. Epub 2011 Dec 15. PMID 22172728
- [Background] Xie X, Atkins E, Lv J, Bennett A, Neal B, Ninomiya T, Woodward M, MacMahon S, Turnbull F, Hillis GS, Chalmers J, Mant J, Salam A, Rahimi K, Perkovic V, Rodgers A. Effects of intensive blood pressure lowering on cardiovascular and renal outcomes: updated systematic review and meta-analysis. Lancet. 2016 Jan 30;387(10017):435-43. doi: 10.1016/S0140-6736(15)00805-3. Epub 2015 Nov 7. PMID 26559744
- [Background] Chowdhury R, Khan H, Heydon E, Shroufi A, Fahimi S, Moore C, Stricker B, Mendis S, Hofman A, Mant J, Franco OH. Adherence to cardiovascular therapy: a meta-analysis of prevalence and clinical consequences. Eur Heart J. 2013 Oct;34(38):2940-8. doi: 10.1093/eurheartj/eht295. Epub 2013 Aug 1. PMID 23907142
- [Background] Roy L, White-Guay B, Dorais M, Dragomir A, Lessard M, Perreault S. Adherence to antihypertensive agents improves risk reduction of end-stage renal disease. Kidney Int. 2013 Sep;84(3):570-7. doi: 10.1038/ki.2013.103. Epub 2013 May 22. PMID 23698228
- [Background] Magacho EJ, Ribeiro LC, Chaoubah A, Bastos MG. Adherence to drug therapy in kidney disease. Braz J Med Biol Res. 2011 Mar;44(3):258-62. doi: 10.1590/s0100-879x2011007500013. Epub 2011 Feb 4. PMID 21344138
- [Background] Karamanidou C, Clatworthy J, Weinman J, Horne R. A systematic review of the prevalence and determinants of nonadherence to phosphate binding medication in patients with end-stage renal disease. BMC Nephrol. 2008 Jan 31;9:2. doi: 10.1186/1471-2369-9-2. PMID 18237373
- [Background] Chang TI, Gao L, Brown TM, Safford MM, Judd SE, McClellan WM, Limdi NA, Muntner P, Winkelmayer WC. Use of secondary prevention medications among adults with reduced kidney function. Clin J Am Soc Nephrol. 2012 Apr;7(4):604-11. doi: 10.2215/CJN.11441111. Epub 2012 Feb 16. PMID 22344513
- [Background] Schmitt KE, Edie CF, Laflam P, Simbartl LA, Thakar CV. Adherence to antihypertensive agents and blood pressure control in chronic kidney disease. Am J Nephrol. 2010;32(6):541-8. doi: 10.1159/000321688. Epub 2010 Nov 2. PMID 21042012
- [Background] Marcum ZA, Sevick MA, Handler SM. Medication nonadherence: a diagnosable and treatable medical condition. JAMA. 2013 May 22;309(20):2105-6. doi: 10.1001/jama.2013.4638. No abstract available. PMID 23695479
- [Background] Crowley MJ, Bosworth HB, Coffman CJ, Lindquist JH, Neary AM, Harris AC, Datta SK, Granger BB, Pereira K, Dolor RJ, Edelman D. Tailored Case Management for Diabetes and Hypertension (TEACH-DM) in a community population: study design and baseline sample characteristics. Contemp Clin Trials. 2013 Sep;36(1):298-306. doi: 10.1016/j.cct.2013.07.010. Epub 2013 Aug 2. PMID 23916915
- [Background] Shrestha SS, Shakya R, Karmacharya BM, Thapa P. Medication adherence to oral hypoglycemic agents among type II diabetic patients and their clinical outcomes with special reference to fasting blood glucose and glycosylated hemoglobin levels. Kathmandu Univ Med J (KUMJ). 2013 Jul-Sep;11(43):226-32. doi: 10.3126/kumj.v11i3.12510. PMID 24442171
- [Background] Nieuwlaat R, Wilczynski N, Navarro T, Hobson N, Jeffery R, Keepanasseril A, Agoritsas T, Mistry N, Iorio A, Jack S, Sivaramalingam B, Iserman E, Mustafa RA, Jedraszewski D, Cotoi C, Haynes RB. Interventions for enhancing medication adherence. Cochrane Database Syst Rev. 2014 Nov 20;2014(11):CD000011. doi: 10.1002/14651858.CD000011.pub4. PMID 25412402
- [Background] Moore SM, Jones L, Alemi F. Family self-tailoring: Applying a systems approach to improving family healthy living behaviors. Nurs Outlook. 2016 Jul-Aug;64(4):306-311. doi: 10.1016/j.outlook.2016.05.006. Epub 2016 May 18. PMID 27301950
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America; Kohn LT, Corrigan JM, Donaldson MS, editors. To Err is Human: Building a Safer Health System. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK225182/ PMID 25077248
- [Background] Russell CL. A clinical nurse specialist-led intervention to enhance medication adherence using the plan-do-check-act cycle for continuous self-improvement. Clin Nurse Spec. 2010 Mar-Apr;24(2):69-75. doi: 10.1097/NUR.0b013e3181cf554d. PMID 20168141
- [Background] Russell CL, Ruppar TM, Matteson M. Improving medication adherence: moving from intention and motivation to a personal systems approach. Nurs Clin North Am. 2011 Sep;46(3):271-81, v. doi: 10.1016/j.cnur.2011.05.004. PMID 21791262
- [Background] Alemi F, Neuhauswer D. A thinking person's step by step guide to changing your lifestyle: Weight loss and exercise program. . Victoria, Canada: Trafford Publishing. 2005.
- [Background] Richard AA, Shea K. Delineation of self-care and associated concepts. J Nurs Scholarsh. 2011 Sep;43(3):255-64. doi: 10.1111/j.1547-5069.2011.01404.x. Epub 2011 Jul 25. PMID 21884371
- [Background] Bronfenbrenner U. Toward an experimental ecology of human development. American psychologist. 1977;32(7):513.
- [Background] Williams A, Manias E, Liew D, Gock H, Gorelik A. Working with CALD groups: testing the feasibility of an intervention to improve medication self- management in people with kidney disease, diabetes, and cardiovascular disease. Renal Society of Australasia
- [Background] Russell CL, Hathaway D, Remy LM, Aholt D, Clark D, Miller C, Ashbaugh C, Wakefield M, Ye S, Staggs VS, Ellis RJ, Goggin K. Improving medication adherence and outcomes in adult kidney transplant patients using a personal systems approach: SystemCHANGE results of the MAGIC randomized clinical trial. Am J Transplant. 2020 Jan;20(1):125-136. doi: 10.1111/ajt.15528. Epub 2019 Aug 20. PMID 31291507
- [Background] Russell C, Conn V, Ashbaugh C, Madsen R, Wakefield M, Webb A, Coffey D, Peace L. Taking immunosuppressive medications effectively (TIMELink): a pilot randomized controlled trial in adult kidney transplant recipients. Clin Transplant. 2011 Nov-Dec;25(6):864-70. doi: 10.1111/j.1399-0012.2010.01358.x. Epub 2010 Nov 16. PMID 21077956
- [Background] Matteson M, Russell C, Winn J. Pilot Intervention to Improve Medication Adherence in Nonadherent Inflammatory Bowel Disease Patients: P-3. Inflammatory Bowel Diseases. 2011;17(Suppl_2):S13-S13.
- [Background] Welch JL, Bartlett Ellis RJ, Perkins SM, Johnson CS, Zimmerman LM, Russell CL, Richards C, Guise DM, Decker BS. Knowledge and Awareness Among Patients with Chronic Kidney Disease Stage 3. Nephrol Nurs J. 2016 Nov-Dec;43(6):513-519. PMID 30550080
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Russell CL, Conn VS, Ashbaugh C, Madsen R, Hayes K, Ross G. Medication adherence patterns in adult renal transplant recipients. Res Nurs Health. 2006 Dec;29(6):521-32. doi: 10.1002/nur.20149. PMID 17131276
- [Background] Radhakrishnan K. The efficacy of tailored interventions for self-management outcomes of type 2 diabetes, hypertension or heart disease: a systematic review. J Adv Nurs. 2012 Mar;68(3):496-510. doi: 10.1111/j.1365-2648.2011.05860.x. Epub 2011 Oct 20. PMID 22010971
- [Background] Finitsis DJ, Pellowski JA, Johnson BT. Text message intervention designs to promote adherence to antiretroviral therapy (ART): a meta-analysis of randomized controlled trials. PLoS One. 2014 Feb 5;9(2):e88166. doi: 10.1371/journal.pone.0088166. eCollection 2014. PMID 24505411
- [Background] Horvath T, Azman H, Kennedy GE, Rutherford GW. Mobile phone text messaging for promoting adherence to antiretroviral therapy in patients with HIV infection. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009756. doi: 10.1002/14651858.CD009756. PMID 22419345
- [Background] Shimohata H, Maruyama H, Ogawa Y, Kobayashi M. Hyperthyroidism associated with obesity-related glomerulopathy-like pathologic features. Intern Med. 2014;53(9):997-9. doi: 10.2169/internalmedicine.53.1814. Epub 2014 May 1. PMID 24785892
- [Background] Callahan CM, Unverzagt FW, Hui SL, Perkins AJ, Hendrie HC. Six-item screener to identify cognitive impairment among potential subjects for clinical research. Med Care. 2002 Sep;40(9):771-81. doi: 10.1097/00005650-200209000-00007. PMID 12218768
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Denhaerynck K, Schafer-Keller P, Young J, Steiger J, Bock A, De Geest S. Examining assumptions regarding valid electronic monitoring of medication therapy: development of a validation framework and its application on a European sample of kidney transplant patients. BMC Med Res Methodol. 2008 Feb 19;8:5. doi: 10.1186/1471-2288-8-5. PMID 18284675
- [Background] Bowling A. Just one question: If one question works, why ask several? J Epidemiol Community Health. 2005 May;59(5):342-5. doi: 10.1136/jech.2004.021204. No abstract available. PMID 15831678
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Result] Bronfenbrenner U. The ecology of human development: Experiments by design and nature. In: Cambridge, MA: Harvard University Press; 1979.
- [Result] Deming E., Orsini J. The Essential Deming: Leadership Principles from the Father of Quality. New York, NY: McGraw-Hill Education; 2012.
- Available data/document: Statistics — https://www.niddk.nih.gov/health-information/health-statistics/kidney-disease — US Department of Health & Human Services. Kidney disease statistics for the United States. Bethesda, MD: National Kidney and Urologic Diseases Information Clearinghouse, National Institutes of Health. 2011.
- Available data/document: Clinical Study Report — https://kdigo.org/wp-content/uploads/2016/10/KDIGO-2012-Blood-Pressure-Guideline-English.pdf — KDIGO. Kidney Disease: Improving global outcomes blood pressure work group, KDIGO clinical practice guideline for the management of blood pressure in chronic kidney disease. Kidney International. 2012;Suppl. 2(5):337-414.
- Available data/document: Clinical Study Report — https://www.niddk.nih.gov/ — National Institute of Diabetes and Digestive and Kidney Diseases. High Blood Pressure and Kidney Disease. In. NIH Publication No. 14-4572 ed. Bethesda, MD: National Kidney and Urologic Diseases Information Clearinghouse (NKUDIC); 2014:12.
- Available data/document: Pamphlet — https://www.nhlbi.nih.gov/resources/brief-your-guide-healthy-sleep-fact-sheet — U.S. Department of Health and Human Services. National Institutes of Health. In Brief: Your Guide to Healthy Sleep. In. Vol NIH Publication No. 11-5800. Bethesda, MA: NHLBI Health Information Center; 2011:1-4.
- Available data/document: Education — https://www.kidney.org/nutrition/Kidney-Disease-Stages-1-4 — National Kidney Foundation. Nutrition and Chronic Kidney Disease (Stages 1-4). Are You Getting What You Need? In. Vol 11-10-1811_HBE. 11-10-1811_HBE ed. New York, NY: National Kidney Foundation; 2013-2014:1-28.
- Available data/document: Education — https://www.kidney.org/atoz/content/Diabetes-and-Kidney-Disease-Stages1-4 — National Kidney Foundation. Hidden health risks: Kidney Disease, Diabetes, and High Blood Pressure. In. Vol 11-10-1811_HBE. New York, NY: National Kidney Foundation 2014:1-20.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded (n = 128)
  * High Adherence (n=53)
  * Lost to follow up (n=41)
  * Change in medication (n=9)
  * Withdrew Consent (n=6)
  * Hospitalization (n=4)
  * Death (n=0)
  * Other (n=15)
    * Cap not received (n=7)
    * Too busy (n=2)
    * Caregiver (n=2)
    * Refused to participate in next phase (n=1)
    * Did not meet inclusion criteria (n=1)
    * Utilizing Pill Packs (n=1)
    * Cap sent back early without communication (n=1)
Groups:
- SystemCHANGE (TM): SystemCHANGE™ focuses on using patients' already established and reliable systems to support medication-taking, rather than focusing on personal effort and "remembering." When applied to medication adherence, the goal is to reduce medication-taking variability and move towards consistently taking medication with a 6-hour window of time (for daily medications like RAAS) and avoid missing medications. SystemCHANGE™ improvement cycles rely on efficient use of performance feedback in order to make decisions about whether system solutions work or if there is a need to select other solutions.
  SystemCHANGE (TM): Participants randomized to the refined SystemCHANGE™ intervention received 7 personalized sessions with a nurse-interventionist (session 1 virtual face-to-face, sessions 2-7 via phone) and 8 weekly feedback MMS message reports delivered to mobile phones.
- Attention Control: Participants in the attention control received educational materials about chronic kidney disease (CKD). The content will be focused on diet, exercise, and stress management with CKD.
  Attention Control: Participants randomized to attention control will receive nurse-led kidney disease self-care education based on materials developed by The National Institute of Diabetes and Digestive and Kidney Diseases and The National Kidney Foundation. Similar to the intervention, participants received 7 personalized sessions with a nurse-interventionist (session 1 virtual face-to-face, sessions 2-7 via phone) and 8 weekly educational MMS messages delivered to mobile phones.
Period: Overall Study
Arm/Group | SystemCHANGE (TM) | Attention Control
Started | 10 | 12
Completed | 4 | 9
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SystemCHANGE (TM) | Attention Control | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 9 | 13
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (9.1) | 59.4 (7.56) | 64.0 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 4 | 2 | 6
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22
Co-morbidities [Count of Participants; unit: Participants]
  Hypertension | 10 | 11 | 21
  Diabetes | 8 | 9 | 17
CKD Stage [Count of Participants; unit: Participants] — During recruitment, collected participant data included stage of chronic kidney disease (CKD), gathered from clinical notes of providing nephrology practitioner. This study was open to those who were in CKD stages 1-4 (better to worse) as defined by kidney disease: Improving global outcomes (KDIGO) and the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) guidelines. CKD is defined as kidney damage where the staging is based on glomerular filtration rate (GFR) range: 1 (normal to high (>90 ml/min/1.73m2) stage 2 (60-89), stage 3a (45-59), 3b (30-44), and stage 4 (15-29).
  Participants
    Stage 1 | 0 | 0 | 0
    Stage 2 | 0 | 2 | 2
    Stage 3a | 4 | 7 | 11
    Stage 3b | 3 | 2 | 5
    Stage 4 | 3 | 1 | 4
CKD etiology [Count of Participants; unit: Participants]
  Diabetes | 0 | 4 | 4
  Hypertension | 3 | 1 | 4
  Not documented | 7 | 5 | 12
  Sickle Cell | 0 | 1 | 1
  Focal segmental glomerulosclerosis (FSGS) | 0 | 1 | 1
Marital Status [Count of Participants; unit: Participants]
  Divorced | 2 | 5 | 7
  Never Married | 3 | 4 | 7
  Married | 2 | 2 | 4
  Widowed | 3 | 1 | 4
Employment Status [Count of Participants; unit: Participants]
  Retired | 7 | 3 | 10
  Disabled | 2 | 4 | 6
  Employed Full Time | 1 | 4 | 5
  Employed Part Time | 0 | 1 | 1
Education [Count of Participants; unit: Participants]
  Less than high school | 1 | 0 | 1
  Some high school | 0 | 2 | 2
  High school graduate | 1 | 3 | 4
  Some college | 3 | 7 | 10
  College Graduate or Higher | 5 | 0 | 5
Income [Count of Participants; unit: Participants]
  Less than $25,000/yr | 5 | 4 | 9
  $25,000 to $50,000/ yr | 0 | 3 | 3
  Over $50,000/yr | 4 | 4 | 8
  Refuse to Answer | 1 | 1 | 2
Insurance Coverage [Count of Participants; unit: Participants]
  Medicare | 5 | 4 | 9
  Medicare plus a supplementary policy | 2 | 0 | 2
  Military/ VA | 0 | 0 | 0
  Medicaid | 3 | 6 | 9
  Private Health Insurance | 1 | 5 | 6
  Don't Know | 1 | 0 | 1
  Other | 1 | 2 | 3
  Refuse to Answer | 0 | 0 | 0
Pill Box Usage [Count of Participants; unit: Participants] — Does participant use a pill box for their medications?
  Participants
    Yes | 5 | 4 | 9
    No | 5 | 8 | 13
Number of Prescribed Daily Medications [Mean (Full Range); unit: Number of Prescribed Medications] | 8.8 [3 to 16] | 10.4 [6 to 21] | 9.7 [3 to 21]
Over the counter medication [Mean (Full Range); unit: Number of OTC Medications] — Average number of over the counter (non-prescription) medications taken on a regular basis within the last three months, such as analgesics, allergy medications, etc.
  (A "regular basis" can be considered medications which are taken more than once per week)
  Number of OTC Medications | 2.5 [0 to 10] | 1.5 [0 to 7] | 2 [0 to 10]
Perceived Health Status [Count of Participants; unit: Participants] — Participants self-rated perceived health
  Participants
    Excellent | 1 | 0 | 1
    Very Good | 1 | 2 | 3
    Good/Fair | 7 | 9 | 16
    Poor | 1 | 1 | 2
    Very Poor | 0 | 0 | 0
Pre-Trial Medication Adherence (8 Weeks-Screening) [Mean (Standard Deviation); unit: Percentage] — Monitored by electronic MEMS caps (AARDEX Group, Belgium) which record the date and time the cap is removed as a proxy for medication being taken. Scale is 0-100%
  Percentage | 83 (9) | 65 (18) | 72 (17)
Systems Thinking Scale [Mean (Standard Deviation); unit: units on a scale] — 20-item Systems Thinking Scale (adapted for patients) was totaled from a 5-point scale (Never, Seldom, Some of the time, Often, Most of the time). Range 20 (personal motivation) -100 (system level thinking). This survey assesses participants view of behavior from a personal (motivation) level to a system (environmental) level. This scale evaluates intervention to improve systems thinking away from a personal motivational thinking. The total score was calculated to evaluate how thinking changed from baseline to 8 weeks and 12 weeks between the groups.
  Dolansky, M. A., et. al (2020). Population: Row population differs as 7 did not complete baseline systems thinking due to lost to follow up before intervention started.
  units on a scale
    number analyzed (Participants) | 6 | 9 | 15
    (all) | 66 (17.06) | 70.92 (17.52) | 70.16 (16.11)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Daily Doses of Medication Taken as Prescribed (Medication Adherence)
Description: Monitored by electronic MEMS caps (AARDEX Group, Belgium) which record the date and time the cap is removed as a proxy for medication being taken.
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: percentage of Daily doses
Arm/Group | SystemCHANGE (TM) | Attention Control
Number analyzed (Participants) | 6 | 8
percentage of Daily doses | 98 (2) | 74 (17)
Statistical Analysis 1: Comparison: SystemCHANGE (TM) vs Attention Control; Test type: Superiority; p = .04, Mixed Models Analysis

2. Primary Outcome: Percentage of Daily Doses of Medication Taken as Prescribed (Medication Adherence)
Description: as for outcome 1
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: percentage of Daily doses
Arm/Group | SystemCHANGE (TM) | Attention Control
Number analyzed (Participants) | 6 | 8
percentage of Daily doses | 91 (9) | 59 (26)
Statistical Analysis 1: Comparison: SystemCHANGE (TM) vs Attention Control; Test type: Superiority; p = .04, ANCOVA

3. Secondary Outcome: Number of Participants Qualitatively Analyzed From the Investigator-designed 10-item Acceptability Questionnaire Which Assesses Nurse-intervention Interaction and Mobile Technology Acceptability.
Description: Response options ranging from 5 (strongly agree) to 1 (strongly disagree). There is no total score. Depending on question "strongly agree" or "strongly disagree" may be related to better acceptability of the intervention. Answers on this survey guided development of individual interview questions to be qualitatively evaluated. The items on the Acceptability Scale, for example, had response options ranging from 5 (strongly agree) to 1 (strongly disagree). If a person indicated strong agreement with the item "Getting messages on the mobile phone helps support my health behaviors," we would develop interview questions to read "You indicated on your survey that getting messages on your phone supported your health behaviors. Tell me what behaviors the messages supported? Give me an example one of these behaviors."
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SystemCHANGE (TM) | Attention Control
Number analyzed (Participants) | 6 | 8
Participants | 6 | 8
Statistical Analysis 1: Comparison: SystemCHANGE (TM) vs Attention Control; Test type: Other; Qualitative data evaluated from interviews tailored after the acceptability scale questionnaire. These interview questions specifically asked participant to rate from strongly disagree to strongly agree on each question and then rationalize answers. Mobile support: 77% of participants agreed that mobile messages supported their health behaviors. Time required: 85% disagreed that the intervention took too much time to learn. Program effectiveness: 92% enjoyed this learning approach, with 100% agreeing they could use the information to improve health behaviors. Rationalization feedback found participants in rural areas reported difficulties accessing texts

4. Secondary Outcome: Outcome Expectancy Questionnaire
Description: This questionnaire measures the affective or emotional aspect of the client's expectations regarding improvement. It asks how much the client expects to improve as a result of the intervention. This is related to the client's emotional responses and affective processes, capturing their hopeful anticipation or optimism about the intervention outcomes.
  Higher scores indicate greater belief that the program will be beneficial. For outcome expectancy, the three questions will indicate how much they 1) think and 2) feel the program will help improve medication-taking using a 0 to 10 scale where 0 is no change and 10 is complete improvement, and how much they 3) feel it will reduce missing or taking medications late using 0 (the intervention won't help to reduce missed doses) to 10 (I won't miss any doses). Responses to the three questions are standardized and summed to create a total subscale score (range 0-30).
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SystemCHANGE (TM) | Attention Control
Number analyzed (Participants) | 6 | 9
score on a scale | 29 (1.3) | 23.7 (5.6)
Statistical Analysis 1: Comparison: SystemCHANGE (TM) vs Attention Control; Test type: Superiority; p = 0.11, Mixed Models Analysis

5. Secondary Outcome: Outcome Expectancy Questionnaire
Description: as for outcome 4
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SystemCHANGE (TM) | Attention Control
Number analyzed (Participants) | 6 | 9
score on a scale | 26.83 (3.13) | 24.57 (7.04)
Statistical Analysis 1: Comparison: SystemCHANGE (TM) vs Attention Control; Test type: Superiority; p = 0.11, Mixed Models Analysis

6. Secondary Outcome: Credibility Questionnaire
Description: This questionnaire measures the logical and cognitive evaluation of the treatment. It assesses how credible or believable the treatment seems to the client. Questions on this scale typically ask about the perceived scientific legitimacy, logic, and reliability of the treatment. It taps into the client's rational thought processes and their cognitive appraisal of the treatment's potential effectiveness.
  Scores on the 3 questions indicate belief the program is credible. For treatment credibility items, participants indicate how 1) logical the program is and 2) how successfully they think it will help prevent missing or taking medications late, and 3) confidence recommending it to a friend all on a 0 to 10 scale and where 0 not logical, not credible, and participant is not confident in recommending to a friend to 10 logical, credible, and would recommend to a friend. Responses are standardized and summed to create a total subscale score on the three questions for a range of 0-30.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SystemCHANGE (TM) | Attention Control
Number analyzed (Participants) | 6 | 9
score on a scale | 28.67 (1.37) | 25.56 (3.50)
Statistical Analysis 1: Comparison: SystemCHANGE (TM) vs Attention Control; Test type: Superiority; p = 0.66, Mixed Models Analysis

7. Secondary Outcome: Credibility Questionnaire
Description: as for outcome 6
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SystemCHANGE (TM) | Attention Control
Number analyzed (Participants) | 6 | 9
score on a scale | 26.67 (4.37) | 25.89 (4.86)
Statistical Analysis 1: Comparison: SystemCHANGE (TM) vs Attention Control; Test type: Superiority; p = 0.66, Mixed Models Analysis

8. Secondary Outcome: Personal Systems Thinking
Description: 20-item Systems Thinking Scale (adapted for patients) was totaled from a 5-point scale (Never, Seldom, Some of the time, Often, Most of the time). Range 20 (personal motivation) -100 (system level thinking). This survey assesses participants view of behavior from a personal (motivation) level to a system (environmental) level. This scale evaluates intervention to improve systems thinking away from a personal motivational thinking. The total score was calculated to evaluate how thinking changed from baseline to 8 weeks and 12 weeks between the groups.
  Dolansky, M. A., et. al (2020).
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SystemCHANGE (TM) | Attention Control
Number analyzed (Participants) | 6 | 8
score on a scale | 68.5 (15.06) | 69.5 (18.51)
Statistical Analysis 1: Comparison: SystemCHANGE (TM) vs Attention Control; Test type: Superiority; p = .84, Mixed Models Analysis

9. Secondary Outcome: Personal Systems Thinking
Description: as for outcome 8
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SystemCHANGE (TM) | Attention Control
Number analyzed (Participants) | 6 | 8
score on a scale | 64.11 (13.27) | 76.17 (15.68)
Statistical Analysis 1: Comparison: SystemCHANGE (TM) vs Attention Control; Test type: Superiority; p = 0.84, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events weekly from 0-8 weeks and then again at 12 weeks.
Arm/Group | SystemCHANGE (TM) | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT04616612/Prot_001.pdf
  • Statistical Analysis Plan (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT04616612/SAP_002.pdf
  • Informed Consent Form (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT04616612/ICF_000.pdf